CLINICAL TRIAL: NCT03107936
Title: Development of a Videogame Prototype Targeting Cigarette and Marijuana Smoking, and Tobacco Product Prevention Among Young Adolescents
Acronym: smokeSCREEN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1401013293
Record Dates: First submitted 2016-12-19; First posted 2017-04-11 (Actual); Last update posted 2018-10-19 (Actual); Status verified 2018-10

CONDITIONS: Smoking
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- smokeSCREEN game play (Experimental): Participants are instructed to access the web-based videogame intervention, smokeSCREEN, through a secured website and play the game using their unique User ID and password.
  Interventions: Behavioral: smokeSCREEN game

INTERVENTIONS:
Behavioral: smokeSCREEN game — smokeSCREEN is web-based videogame intervention focused on tobacco use prevention in teens. The game has 1.5-2 hours of unique game play and focuses on combustible cigarettes, e-cigarettes, and flavored tobacco products.smokeSCREEN. Guided by the social cognitive theory and the theory of planned behavior, smokeSCREEN addresses a range of challenges that teens often face involving peer pressure and the use of tobacco products. Participants are provided access to the smokeSCREEN game through a private, password-protected website link and instructed to complete the game.

SUMMARY:
To study feasibility and implementation of a education videogame and the effects on adolescents knowledge and beliefs around tobacco products.

DETAILED DESCRIPTION:
The goal for sub-study 4 is to learn more about how an educational videogame can feasibly be implemented and disseminated in youth programs. For this sub-study we will further develop, expand, and refine the smokeSCREEN game and increase the game's reach on a national platform. The study will conduct the proposed evaluation by: working with game developers to develop a web- based version of the game, creating a pre-post survey to measure the effect of the game and building that into the smokeSCREEN game to anonymously collect information on players' knowledge and beliefs around tobacco products, and collaborating with youth programs to pilot test how the game can be implemented in real world settings.

ELIGIBILITY:
Inclusion Criteria:

* must be able and willing to sit at a computer or mobile device for 45-60 minutes per session to play the game and answer questions before and after playing video game.
* be enrolled in a youth program that we have a partnership with

Exclusion Criteria:

* up to the discretion of the study team

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Beliefs about smoking pre-test survey | Baseline
  Participants completed a pre-survey through a secured, data collection website (Qualtrics Data Collection Software) and then played the videogame intervention. Fourteen questions were designed from the National Youth Tobacco Survey (2014)13 that focused on beliefs about cigarettes, e-cigarettes, and flavored tobacco were used. For beliefs, questions had 4-5 choices ranging from strongly disagree to strongly agree or definitely yes to definitely not, or 5 response choices ranging from very unlikely to very likely.
Beliefs about smoking post-test survey | immediately after game play is completed
  Participants completed a post-survey through a secured, data collection website (Qualtrics Data Collection Software), after they have played the videogame intervention. Fourteen questions were designed from the National Youth Tobacco Survey (2014)13 that focused on beliefs about cigarettes, e-cigarettes, and flavored tobacco were used for the survey. For beliefs, questions had 4-5 choices ranging from strongly disagree to strongly agree or definitely yes to definitely not, or 5 response choices ranging from very unlikely to very likely.
Knowledge about smoking pre-test survey | Baseline
  Participants completed a pre-survey through a secured, data collection website (Qualtrics Data Collection Software), played the videogame intervention. Fourteen questions were designed from the National Youth Tobacco Survey (2014)13 that focused on knowledge about cigarettes, e-cigarettes, and flavored tobacco were used for the surveys. For knowledge, questions had 3 response choices (yes, not, and not sure).
Knowledge about smoking post-test survey. | immediately after game play is completed
  Participants completed a pre-survey through a secured, data collection website (Qualtrics Data Collection Software), played the videogame intervention, and then completed a post-survey using the same data collection website. Fourteen questions were designed from the National Youth Tobacco Survey (2014)13 that focused on knowledge about cigarettes, e-cigarettes, and flavored tobacco were used for the survey. For knowledge, questions had 3 response choices (yes, not, and not sure).
Game experience satisfaction post-test survey | immediately after game play is completed
  The post-test survey included an additional 5 items on game experience and satisfaction from items designed for a previous videogame study on sexual risk reduction in young adolescents (e.g., "I would tell my friends to play this game," 4 response choices, ranging from strongly disagree to strongly agree).

CONTACTS AND LOCATIONS:
Overall Officials: Lynn E. Fiellin, MD, Principal Investigator — Yale University
Locations (4):
- United States (4):
  - Hamden Youth Center, Hamden, Connecticut
  - Leadership, Education, and Athletics Partnership (LEAP) Inc., New Haven, Connecticut
  - Yale New Haven Hospital, New Haven, Connecticut
  - Farnam Neighborhood House, New Haven, Connecticut

IPD SHARING:
Plan to Share IPD: No